CLINICAL TRIAL: NCT06867055
Title: Evaluation of the Efficacy of Injectable Platelet Rich Fibrin (I-TZF) Impregnated Gelatin Sponge and 0.8% Hyaluronic Acid Gel Impregnated Gelatin Sponge on Clinical Healing of Palatinal Wound Healing After Free Gingival Grafting.
Brief Title: Evaluation of the Effectiveness of Different Procedures on Palatinal Wound Healing After Free Gingival Graft Surgery.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, SEVAL CEYLAN ŞEN, Assist Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Seval1
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Insufficient Keratinized Gingiva
Keywords: wound healing; analog pain scale; free gingival graft; injectable plathelet rich fibrin; palate; Wound epithelization; topical hyaluronic acid
MeSH Terms: interventions — proliferation regulatory factors, human urine; Control Groups

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, single blind, parallel group controlled clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I-PRF (Experimental): ]. In the first test group, based on the g force, peripheral blood was collected in sterile plain plastic tubes (Beliver Industrial Estate, Pylmouth, UK.) and centrifuged to obtain I-PRF [16]. Injectable platelet-rich fibrin was produced using a protocol of 2500 RPM for 3 min (RCF-max = 509.53 g) I-PRF were produced with 11-mL plastic tubes (16*10 mm) using a Nuve NF 200 centrifugation device with a rotor angulation with a radius of 101 mm at the clot (Nuve NF 200, Nuve Industrial Materials Manufacturing and Trade Company, Ankara, Türkiye). The I-PRF at the top of the tube was collected with a syringe and transferred to the metal bowl. It was held for 20-25 min for polymerization. In the I-PRF test group, I-PRF was impregnated on a sterile gelatin sponge and sutured with 4/0 silk suture (4/0 Sterisilk, SSM Medical Equipment, Türkiye) on the palate area and bleeding was controlled with SX bioplast plate.
  Interventions: Biological: Injectable platelet-rich fibrin (I-PRF)
- Gengigel (HA) (Experimental): 0.8% polyvinylpyrrolidone sodium hyaluronate (HA) (Gengigel Prof, Ricerfarma SRL.) gel was impregnated on a sterile gelatin sponge and sutured with 4/0 silk suture (4/0 Sterisilk, SSM Medical Equipment, Türkiye) on the palate area and bleeding control was provided with SX bioplast plate.
  Interventions: Drug: 0.8% hyaluronic acide (HA)
- Control (Experimental): Only sterile gelatin sponge was sutured with 4/0 silk suture (4/0 Sterisilk, SSM Medical Equipment, Turkey) in the palatal region where FGG was taken and bleeding was controlled with SX bioplast plate.
  Interventions: Other: control group

INTERVENTIONS:
Biological: Injectable platelet-rich fibrin (I-PRF) — I-PRF were produced with 11-mL plastic tubes (16*10 mm) using a Nuve NF 200 centrifugation device with a rotor angulation with a radius of 101 mm at the clot (Nuve NF 200, Nuve Industrial Materials Manufacturing and Trade Company, Ankara, Türkiye). The I-PRF at the top of the tube was collected with a syringe and transferred to the metal bowl. It was held for 20-25 min for polymerization.
  Arms: I-PRF
Drug: 0.8% hyaluronic acide (HA) — 0.8% polyvinylpyrrolidone sodium hyaluronate (HA) (Gengigel Prof, Ricerfarma SRL.) gel was impregnated on a sterile gelatin sponge and sutured with 4/0 silk suture (4/0 Sterisilk, SSM Medical Equipment, Türkiye) on the palate area and bleeding control was provided with SX bioplast plate.
  Arms: Gengigel (HA)
Other: control group — Sterile gelatin sponge was sutured with 4/0 silk suture (4/0 Sterisilk, SSM Medical Equipment, Turkey) in the palatal region where FGG was taken and bleeding was controlled with SX bioplast plate.
  Arms: Control

SUMMARY:
This study aimed to help determine the appropriate method to accelerate wound healing at the free gingival graft donor site and to minimize the patient's postoperative complaints. For this purpose, gelatin sponge impregnated with injectable platelet-rich fibrin (I-PRF), gelatin sponge impregnated with 0.8% polyvinylpyrrolidone sodium hyaluronate (HA) gel, and standard gelatin sponge application were compared to the secondary wound site on the palate.

The main questions aimed at being answered are:

* Does the use of I-PRF or HA accelerate wound healing in patients?
* Does the use of I-PRF or HA reduce pain and burning symptoms?
* For this purpose, gelatin sponge impregnated with injectable platelet-rich fibrin (I-PRF), gelatin sponge impregnated with 0.8% polyvinylpyrrolidone sodium hyaluronate (HA) gel, and standard gelatin sponge application were compared to the secondary wound site on the palate.

Participants will:

* They will record whether there is pain and burning for 7 days after the operation.
* They will record if there is bleeding in the palate area.
* They will write the number of painkillers they use daily.
* They will visit the clinic on the 3rd, 5th, 7th, 14th, 21st, 28th days and 1st and 3rd months after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study were;
* patients older than 18 and
* systemically healthy patients,
* who didn't use drugs that affect wound healing,
* didn't have coagulation disorder and nausea, and
* were not anti-inflammatory drug allergy sufferers.

Exclusion Criteria:

* Exclusion criteria for the study were;
* patients who had systematic disorders (such as diabetes, hypertension, radiotherapy, chemotherapy),
* patients who were former or active smokers and alcohol users,
* pregnant and breastfeeding, lactation, menstruation,
* patients with poor oral hygiene, and patients who didn't attend regular check-ups.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Landry Wound Healing Index (WHI) | 1st, 3rd, 7th, 14th, 21st, 28th days and 1st and 3rd month after the surgical procedure
  The primary result expected from the study is that the healing of the palatinal region left for secondary healing is faster in the I-PRF and 0.8% HA groups compared to the control group.
  The primary outcome of the study was to measure the palatal wound healing status using the Landry Wound Healing Index (WHI) (Landry RG (1985) Efectiveness of benzydamine HC1 in the treatment of periodontal post-surgical patients. Faculty of Dentistry, University of Toronto), which grades the wound healing on a scale of the 3rd, 7th, 14th, 21st, and 28th days postoperatively. This index, which has a score range of 1 (very poor) to 5 (excellent), evaluates tissue color, response to palpation, granulation tissue presence, incision margins' epithelialization, and amount of suppuration.

SECONDARY OUTCOMES:
pain and burn (Visual Analog Scale) | First 7 day after the surgical procedure
  The secondary result expected from the study is that postoperative pain and burning are less in the I-PRF and 0.8% HA groups compared to the control group.
  The secondary outcomes of the study were to measure patients' perception of pain, discomfort while chewing, and burning sensation after FGG harvesting using a numerical rating scale (VAS) from 0 (no pain, no discomfort while chewing, no burning sense) to 10 (the worst pain imaginable, extreme discomfort while chewing, extreme burning sense) between days 1 and 7, and the amount of analgesic consumption between days 1 and 7 postoperatively.
Tissue color match (CM) | 1st, 3rd, 7th, 14th, 21st, 28th days and 1st and 3rd month after the surgical procedure
  Tissue color match (CM) was assessed with adjacent and contralateral palatal tissue (0-no color matching to 10-excellent color matching)
postoperative bleeding | 1st, 3rd, 5th, and 7th day after the surgical procedure.
  The patients were asked to keep a record of whether there was any bleeding in the palatal region, and at the same time, the presence of postoperative bleeding, also known as delayed bleeding (DB), was recorded as present (+) or absent (-) on the days when the patients came to the follow up appointments.
H2O2 bubbling | 1st, 3rd, 7th, 14th, 21st, 28th days after the surgical procedure
  The epithelialization of the palatal region was recorded according to the application of 3% hydrogen peroxide to the region and whether there was foaming or not, and was calculated as a percentage (H2O2 bubbling). Complete epithelization (CE) was also evaluated clinically by monitoring the surface characteristics and clarity of the wound contour and recorded as "yes" or "no".
Oral Health Related Quality of Life (OHRQoL) | 7th and 14th days after the surgical procedure.
  Oral Health Related Quality of Life (OHRQoL) was administered on the 7th and 14th days after the surgical procedures to analyse how the person's daily physical-social life and mental health status were affected. This scale developed by McGrath and Bedi evaluates the effects of oral health on quality of life in both positive and negative domains. The scale includes 16 questions consisting of 4 different categories. The categories consist of current symptoms (2 questions) and physical (5 questions), psychological (5 questions) and social (4 questions) conditions. The questions in the OHRQOL-TR questionnaire are scored on a Likert scale with values between 1 and 5 (such as 'very bad' (score 1), 'bad' (score 2), 'none' (score 3), 'good' (score 4) or 'very good' (score 5)). When the scores of 16 questions are totalled, there is a value in the range of 16-80. The reliability and validity of the Turkish version of the scale was proved and reported in the study conducted by Mumcu et al.
Number of analgesics taken | First 7 day after the surgical procedure.
  Patients were informed that the number of analgesics theytook for post-operative pain relief was recorded for 7 days
palatal soft-tissue thickness (PSTT) | Initial, 1st and 3rd month after the surgical procedure
  The PSTT in the harvested area was measured after theadministration of local anaesthesia.The measurement was made approximately 5 mm apical to the gingival marginof the first premolar using a #15 endodontic reamer. Thepenetration depth was measured using a digital caliper. Themeasurements were obtained before harvesting the FGG and at 1 and 3 months after the operation.The graft thickness was measured in the same way at the middle points of all four edges of the graft. The mean of theobtained values was calculated and considered to be the graft thickness. The dimensions of the graft were standardized using a sterile aluminium foil template of 7 * 12 mm.
tissue consistency | On the 3rd, 7th, 14th and 21st days after surgery
  After the operation, the consistency of the donor area in the palatal region was marked to be soft and firm.
Palate sensitivity | On the 7th, 14th and 21st days after surgery
  Palate sensitivity was measured by using a numerical rating scale (VAS) from 0 (no sensitivity) to 10 (most sensitivity) on the 7th, 14th and 21st days after surgery
Loss of sensation | n the 3rd, 7th, 14th, 21st, 28th day, 1st month, and 3rd month after the operation
  Loss of sensation was recorded as none (0), moderate (1), and severe (2) on the 3rd, 7th, 14th, 21st, 28th day, 1st month, and 3rd month after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: SEVAL CEYLAN ŞEN, Assist Prof., Principal Investigator — Gülhane Diş Hekimliği Fakültesi
Locations (1):
- Health Sciences University Gulhane Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceylan Sen S, Sarac Atagun O, Ustaoglu G, Ozcan E. Comparative evaluation of hyaluronic acid and injectable platelet-rich fibrin in palatal wound healing: a randomized clinical trial. BMC Oral Health. 2025 Oct 29;25(1):1693. doi: 10.1186/s12903-025-07183-9. PMID 41162972